CLINICAL TRIAL: NCT00867269
Title: Etiology, Pathogenesis, and Natural History of Idiopathic CD4+ Lymphocytopenia
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090102; 09-I-0102
Record Dates: First submitted 2009-03-20; First posted 2009-03-23 (Estimated); Last update posted 2026-01-12 (Actual); Status verified 2026-01-08

CONDITIONS: Idiopathic CD4+ Lymphocytopenia; Cryptococcal Meningitis; Warts
Keywords: Opportunistic Infection; Immunodeficiency Syndrome; Autoimmune Disease; CD4+ Lymphocytes; Natural History; Idiopathic CD4 Lymphocytopenia
MeSH Terms: conditions — T-Lymphocytopenia, Idiopathic CD4-Positive; Meningitis, Cryptococcal; Warts; Opportunistic Infections; Immunologic Deficiency Syndromes; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Blood Relatives: Blood Relatives of ICL subjects
- Household Contacts: Household contacts of ICL subjects
- ICL Subjects: Patients with confirmed idiopathic CD4 lymphocytopenia

SUMMARY:
Background:

* Idiopathic CD4+ lymphocytopenia (ICL) is a condition in which there is a decreased level of CD4+ lymphocytes (a type of white blood cell), which can lead to opportunistic infections or autoimmune disorders and diseases.

Objectives:

* To characterize the natural history with regard to CD4+ T cell count and onset of infection, malignancy, and autoimmunity.
* To describe the immunological status of patients affected by ICL while providing the best possible standard therapy to eradicate opportunistic infections.
* To establish the timeline of CD4 lymphocytopenia, with particular focus on defining subgroups of patients according to the decline, stabilization, or rise of CD4+ T cell counts over time.
* To characterize the opportunistic infections that occur in ICL patients at microbiologic and molecular levels.
* To characterize the immunophenotype and possible genetic immunodeficiency causes of ICL.
* To determine whether measurable immunologic parameters correlate with the development of opportunistic infections or other comorbidities such as lymphoma in patients with ICL.
* To determine whether there is any association between ICL and autoimmunity.
* To determine CD4+ T cell turnover, survival, functionality, and cytokine responsiveness in ICL patients.

Eligibility:

* Patients 2 years of age and older with an absolute CD4 count less than 300 in children 6 years or older and adults or less than 20% of T cells in children younger than 6 on two occasions at least 6 weeks apart.
* Patients with negative results of HIV testing by ELISA, Western Blot, and viral load.
* Patients must not have underlying immunodeficiency conditions, be receiving cytotoxic chemotherapy (anti-cancer drugs that kill cells), or have cancer.

Design:

* At the initial visit to the National Institutes of Health, the following evaluations will be conducted:
* Personal and family medical histories.
* Physical examination, including rheumatology evaluation and other consultations as medically indicated (e.g., dermatology, pulmonology, ophthalmology, imaging studies).
* Blood samples for analysis of red and white blood cell counts, liver function, immune hormones, and antibody and autoantibody levels, white blood cell growth and function, and DNA.
* Urinalysis and urine pregnancy testing for female patients of childbearing age.
* Evaluation and treatment of active infections as medically indicated, including biopsies, buccal swabs, pulmonary function tests, and imaging studies.
* Follow-up visits will take place approximately every 12 months or more frequently if indicated, and will continue for a minimum of 4 years and a maximum of 10 years.
* Evaluations at follow-up will include blood samples (i.e., CBC with differential, biochemical profile, HIV testing, etc.) and urinalysis and rheumatology consults.

DETAILED DESCRIPTION:
Idiopathic CD4+ lymphocytopenia (ICL) is a disorder characterized by decreased numbers of circulating CD4+ T lymphocytes in the absence of known causes of CD4+ lymphocytopenia. ICL is defined as an absolute CD4+ T cell count of less than 300 cells/microL in a patient with no human immunodeficiency virus infection or known immunodeficiency syndrome. The causes and frequency of the disorder remain unknown. The condition is typically diagnosed when patients present with a serious infection. In this natural history protocol, we will evaluate patients with CD4+ T cell counts below 300 cells/microL. We propose to follow 300 ICL patients for a minimum of 4 and maximum of 20 years, with a particular focus on the association between ICL and autoimmune disease. In addition to the ICL patients, we will enroll blood relatives and household contacts to better understand pathogenesis and etiologies of the syndrome. We will collect blood and other tissues for immunologic, rheumatologic, and genetic testing in an effort to identify and understand the underlying defects that cause ICL and follow its course in a cohort of patients who will receive best standard therapy for opportunistic infections.

ELIGIBILITY:
* ICL PARTICPANT INCLUSION CRITERIA:

To be eligible for this study, patients must satisfy all of the following inclusion criteria:

1. Age greater than or equal to 18 years
2. Absolute CD4 count < 300 cells/microL or < 20% of total T cells on at least two occasions at least 6 weeks apart
3. Ongoing care by a referring primary care physician
4. Willingness to allow storage of blood and tissue samples for future analysis

ICL PARTICPANT EXCLUSION CRITERIA:

Patients will be ineligible for this study if they satisfy any of the following criteria:

1. Known infection with HIV-1, HIV-2, or human T-cell lymphotropic viruses (HTLV-1 or HTLV-2) as demonstrated by enzyme-linked immunosorbent assay (ELISA) and western blot and/or viral load testing
2. Known underlying immunodeficiency syndrome other than ICL
3. Evidence of active malignancy
4. Receipt of medications, herbal substances, or biologic agents known to diminish the CD4+ count within 30 days of when the CD4+ lymphocytopenia was detected
5. Any condition that in the judgment of the investigators would place the subject at undue risk or compromise the results of the study.

BLOOD RELATIVE INCLUSION CRITERIA:

To be eligible for study participation as a blood relative, subjects must be greater than or equal to 18 years of age and be a blood relative of an individual who meets or has met the CDC criteria for ICL.

HOUSEHOLD CONTACT INCLUSION CRITERIA:

To be eligible for study participation as a household contact, subjects must be greater than or equal to18 years of age and live within the same household as an ICL subjects participating in this protocol. Blood relatives who are household contacts are eligible to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with idiopathic CD4+ lymphocytopenia (ICL) who have CD4 <300/microliters or < 20% of total T cells and their blood relatives and household contacts.
Sampling Method: Non-Probability Sample
Enrollment: 950 (Estimated)
Dates: Start 2009-07-13 (Actual)

PRIMARY OUTCOMES:
CD4 <300/microliters or < 20% of total T cells and their blood | Baseline and annually
  To further characterize the natural history of ICL while also investigating the genetic, environmental, and immunologic features of the condition.

SECONDARY OUTCOMES:
Determine CD4+ T cell turnover, survival, functionality and cytokineresponsiveness in selected ICL patients. | Baseline and annually
  Collection of research blood (PBL, serum and plasma) for storage
Investigate ICL immune cell homeostasis and trafficking by immunologic studies including tissue biopsies and the utilization of ahumanized mouse model. | Baseline and annually
  Collection of research blood (PBL, serum and plasma) for storage
Establish the prognosis of CD4 lymphocytopenia, with particular focus on defining subgroups of patients according to the decline, stabilization, or rise of CD4+T cell counts over time. | Baseline and annually
  Collection of research blood (PBL, serum and plasma) for storage
Determine whether measurable immunologic parameters correlate with the development of opportunistic infections or other co-morbidities | Baseline and annually
  Determine whether measurable immunologic parameters correlate with the development of opportunistic infections or other co-morbidities such as lymphoma in patients with ICL. Investigate the associations between idiopathic CD4+ lymphocytopenia and autoimmunity.Collection of research blood (PBL, serum and plasma) for storage
Determine the relationship between ICL and the microbiome. | Baseline and annually
  Collection of rectal swab and dietary questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Irini Sereti, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Fauci AS. CD4+ T-lymphocytopenia without HIV infection--no lights, no camera, just facts. N Engl J Med. 1993 Feb 11;328(6):429-31. doi: 10.1056/NEJM199302113280610. No abstract available. PMID 8093637
- [Background] Laurence J, Siegal FP, Schattner E, Gelman IH, Morse S. Acquired immunodeficiency without evidence of infection with human immunodeficiency virus types 1 and 2. Lancet. 1992 Aug 1;340(8814):273-4. doi: 10.1016/0140-6736(92)92359-n. PMID 1353194
- [Background] Ho DD, Cao Y, Zhu T, Farthing C, Wang N, Gu G, Schooley RT, Daar ES. Idiopathic CD4+ T-lymphocytopenia--immunodeficiency without evidence of HIV infection. N Engl J Med. 1993 Feb 11;328(6):380-5. doi: 10.1056/NEJM199302113280602. PMID 8093634
- [Derived] Lisco A, Ortega-Villa AM, Mystakelis H, Anderson MV, Mateja A, Laidlaw E, Manion M, Roby G, Higgins J, Kuriakose S, Walkiewicz MA, Similuk M, Leiding JW, Freeman AF, Sheikh V, Sereti I. Reappraisal of Idiopathic CD4 Lymphocytopenia at 30 Years. N Engl J Med. 2023 May 4;388(18):1680-1691. doi: 10.1056/NEJMoa2202348. PMID 37133586
- [Derived] Sortino O, Dias J, Anderson M, Laidlaw E, Leeansyah E, Lisco A, Sheikh V, Sandberg JK, Sereti I. Preserved Mucosal-Associated Invariant T-Cell Numbers and Function in Idiopathic CD4 Lymphocytopenia. J Infect Dis. 2021 Aug 16;224(4):715-725. doi: 10.1093/infdis/jiaa782. PMID 34398238
- [Derived] Perez-Diez A, Wong CS, Liu X, Mystakelis H, Song J, Lu Y, Sheikh V, Bourgeois JS, Lisco A, Laidlaw E, Cudrici C, Zhu C, Li QZ, Freeman AF, Williamson PR, Anderson M, Roby G, Tsang JS, Siegel R, Sereti I. Prevalence and pathogenicity of autoantibodies in patients with idiopathic CD4 lymphopenia. J Clin Invest. 2020 Oct 1;130(10):5326-5337. doi: 10.1172/JCI136254. PMID 32634122
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2009-I-0102.html